CLINICAL TRIAL: NCT00456222
Title: Impact of Sleep Disruption on the Menstrual Cycle
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Elizabeth B. Klerman, MD, PhD, Brigham & Women's Hospital
Other Study IDs: R01HD040291 (NIH); NIH R01-HD40291
Record Dates: First submitted 2007-04-02; First posted 2007-04-04 (Estimated); Last update posted 2009-08-21 (Estimated); Status verified 2009-08

CONDITIONS: Sleep; Circadian Rhythm; Menstrual Cycle
Keywords: Sleep; Circadian rhythms; Menstrual cycle

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood/plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Luteal
  Interventions: Behavioral: Disrupting or changing the timing or the duration of sleep
- Follicular
  Interventions: Behavioral: Disrupting or changing the timing or the duration of sleep

INTERVENTIONS:
Behavioral: Disrupting or changing the timing or the duration of sleep — Disrupting or changing the timing or the duration of sleep

SUMMARY:
The purpose of this study is to investigate whether sleep disruption affects menstrual cycle timing

DETAILED DESCRIPTION:
Menstrual cycle dynamics were studied after sleep disruption

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Regular menstrual cycles

Exclusion Criteria:

* No medications affecting the menstrual cycle or sleep

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy women with regular menstrual cycles
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2003-06; Primary Completion 2007-07 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth B Klerman, MD PhD, Principal Investigator — Brigham and Women's Hospital; Janet E Hall, MD, Study Director — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts